CLINICAL TRIAL: NCT03312491
Title: Treatment of Acetabular Fracture: the Contribution of the 3D Impression
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 3D COTYLE
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetabular fracture are common in elder patients and high energy trauma in younger one.

However, the fracture deplacement induces incongruity between cotyloid cavity and femoral head. Anatomic reduction and osteosynthesis of these fracture are technically difficult .

3D printing ease the process of operating planification or implant fabrication. The 3D impression allows to obtain a model on the scale of the pond of the patient allowing to pre mold plates on the anatomy of the patient before he is operated with the aim of decreasing the surgical time and improving the quality of the reduction.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* acetabulum fracture within one month
* anterior access or double access

Exclusion Criteria:

* acetabulum fracture more than one month

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient admitted in orthopaedic yard for acetabulum fracture
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
operating room time | day1

CONTACTS AND LOCATIONS:
Overall Officials: Pomme JOUFFROY, MD, Study Chair — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France